CLINICAL TRIAL: NCT01706666
Title: A Phase II Randomized Study of Three Subcutaneous Bortezomib-based Consolidation Treatments for Patients Completing Induction Therapy and Stem Cell Transplantation for Newly Diagnosed Multiple Myeloma
Brief Title: Bortezomib Based Consolidation in Multiple Myeloma Patients Completing Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1186; NCI-2012-01579 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-08

CONDITIONS: Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
Keywords: Maintenance; Consolidation
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclophosphamide; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (bortezomib) (Experimental): Patients receive bortezomib SC on days 1 and 15 of courses 1-12 and day 1 of courses 13-24.
  Interventions: Drug: bortezomib; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment
- Arm B (bortezomib, cyclophosphamide, dexamethasone) (Experimental): Patients receive bortezomib SC as in Arm A, cyclophosphamide PO on days 1 and 15 of courses 1-12 and day 1 of courses 13-24, and dexamethasone PO on days 1 and 15 of courses 1-12 and day 1 of courses 13-24.
  Interventions: Drug: bortezomib; Drug: cyclophosphamide; Other: laboratory biomarker analysis; Drug: dexamethasone; Procedure: quality-of-life assessment
- Arm C (bortezomib, lenalidomide) (Experimental): Patients receive bortezomib SC as in Arm A and lenalidomide PO QD on days 1-28.
  Interventions: Drug: bortezomib; Drug: lenalidomide; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: bortezomib — Given SC
  Other Names: LDP 341; MLN341; VELCADE
Drug: cyclophosphamide — Given PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Arm B (bortezomib, cyclophosphamide, dexamethasone)
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
  Arms: Arm C (bortezomib, lenalidomide)
Other: laboratory biomarker analysis — Correlative studies
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
  Arms: Arm B (bortezomib, cyclophosphamide, dexamethasone)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized phase II trial studies how well giving bortezomib with or without combination chemotherapy works as consolidation therapy in patients with newly diagnosed multiple myeloma who have completed stem cell transplant. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide, dexamethasone, and lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving bortezomib is more effective with or without combination chemotherapy in the post transplant setting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the stringent complete response (sCR) rate after 12 cycles among arms.

SECONDARY OBJECTIVES:

I. To compare progression-free and overall survival among arms. II. To describe the adverse event profile of each arm.

TERTIARY OBJECTIVES:

I. To compare sCR after 6 cycles and 24 cycles and quality of life among arms.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A: Patients receive bortezomib subcutaneously (SC) on days 1 and 15 of courses 1-12 and day 1 of courses 13-24.

ARM B: Patients receive bortezomib SC as in Arm A, cyclophosphamide orally (PO) on days 1 and 15 of courses 1-12 and day 1 of courses 13-24, and dexamethasone PO on days 1 and 15 of courses 1-12 and day 1 of courses 13-24.

ARM C: Patients receive bortezomib SC as in Arm A and lenalidomide PO once daily (QD) on days 1-28.

In all arms, treatment continues every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Creatinine =< 2 mg/dL
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 75000/mm^3
* Hemoglobin >= 8.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Treated myeloma: Prior induction therapy (any) and followed by autologous stem cell transplantation
* Measurable disease at initial diagnosis, pre-stem cell transplant (SCT) or post-SCT of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 0.5 g/dL
  * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 5 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis >= 30% (evaluable disease)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* < 120 days post SCT with no evidence of relapse or progression prior to registration
* Provide voluntary informed written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to return to enrolling institution for follow-up during the active monitoring phase of the study
* Ability to complete questionnaire(s) by themselves or with assistance
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study treatment, OR agree to completely abstain from heterosexual intercourse
* Male patients, even if surgically sterilized (ie, status postvasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study treatment, OR
  * Agree to completely abstain from heterosexual intercourse

Exclusion Criteria:

* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Known to be human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus positive (HBV+)
* Hypersensitivity to study drugs, boron or mannitol
* Patient refractory to bortezomib (defined as patients who progressed while on bortezomib or within 60 days of receiving bortezomib)
* Any serious medical or psychiatric condition that would prevent the subject from complying with the protocol treatment and procedures
* Grade >= 2 peripheral neuropathy
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial
* Radiation therapy within 3 weeks before randomization; enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy
* Female patients who are lactating or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2014-07-10 (Actual); Study Completion 2016-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig B. Reeder, M.D., Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Baylor Medical Center, Garland, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Patients receive bortezomib SC on days 1 and 15 of courses 1-12 and day 1 of courses 13-24.
- Arm B: Patients receive bortezomib SC as in Arm A, cyclophosphamide PO on days 1 and 15 of courses 1-12 and day 1 of courses 13-24, and dexamethasone PO on days 1 and 15 of courses 1-12 and day 1 of courses 13-24.
- Arm C: Patients receive bortezomib SC as in Arm A and lenalidomide PO QD on days 1-28.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 1 | 1 | 1
Completed | 1 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Continuous [Median (Full Range); unit: Years] | 54 | 45 | 50 | 50 [45 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 1 | 0 | 1 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 3
Had Prior Treatment [Number; unit: participants] | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Experiencing a Stringent Complete Response (sCR) After 12 Cycles, 24 Months
Description: Estimated by the number of sCRs divided by the total number of evaluable patients in each arm. Exact binomial confidence intervals for the true sCR rate will be calculated by arm. Stringent complete response (sCR) is defined as a complete response plus normal serum free light chain ratio and the absence of clonal cells in bone marrow by flow cytometry.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 1 | 1 | 1
percentage of participants | 100 | 0 | 100

2. Secondary Outcome: Survival Time
Description: The distribution of survival time will be estimated by arm using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, assessed up to 3 years
Population: All patients are still alive
Measure: Number; unit: Months to death
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 1 | 1 | 1
Months to death | NA — No Deaths | NA — No Deaths | NA — No Deaths

3. Secondary Outcome: Progression-free Survival
Description: The distribution of progression-free survival will be estimated by arm using the method of Kaplan-Meier.
Time Frame: From registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 3 years
Measure: Number; unit: Months to Progression
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 1 | 1 | 1
Months to Progression | NA — No progressions | 9.2 | NA — No progressions

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B | Arm C
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=1) | Arm B (N=1) | Arm C (N=1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=1) | Arm B (N=1) | Arm C (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (5) | 1 (10) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (10)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (7) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (9) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (6) | 1 (13)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (10)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (10)
White blood cell decreased (Investigations) | 0 (0) | 1 (5) | 1 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes